CLINICAL TRIAL: NCT00549406
Title: Visual Processing and Postural Reactions: Development and Pilot Testing of a "Visual Training" Program to Improve Balance Control and Prevent Falls in Older Adults
Brief Title: Visual Training Program to Improve Balance and Prevent Falls in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Neurotrauma Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr Brian Maki, Director, Centre for Studies in Aging, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-PREV-INT-452; CIHR grant# MOP-13355
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Accidental Falls; Musculoskeletal Equilibrium
Keywords: Vision; Visual attention; Postural balance; Geriatrics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): computer-based visual-training program UFOV
  Interventions: Procedure: computerized visual training
- 2 (Experimental): video-game based visual training
  Interventions: Procedure: video-game based visual training
- 3 (Placebo Comparator): computerized word puzzles
  Interventions: Procedure: computerized word puzzles

INTERVENTIONS:
Procedure: computerized visual training — two one-hour training sessions per week, for five consecutive weeks
  Other Names: "Useful Field of View" (UFOV) training
  Arms: 1
Procedure: computerized word puzzles — two one-hour sessions per week, for five consecutive weeks
  Other Names: "Super Text-Twist" puzzles
  Arms: 3
Procedure: video-game based visual training — two one-hour training sessions per week, for five consecutive weeks
  Other Names: Video game training
  Arms: 2

SUMMARY:
The ability to maintain balance and avoid falling is highly dependent on the ability to locate objects and architectural features in the environment. This need to continually monitor the environment as one moves about in daily life suggests a critical role for visual attention, gaze control, and spatial memory, all of which are known to decline with aging. In this study, the investigators will test the efficacy of a computer-based visual-training program designed to improve the ability to rapidly extract information from the peripheral visual field. It is expected that older adults involved in the visual training intervention will improve the speed, accuracy, and effectiveness of reach-to-grasp balance-recovery reactions evoked by sudden unpredictable balance perturbation.

DETAILED DESCRIPTION:
Balance reactions that involve rapidly stepping or reaching to grasp a handrail or other objects for support play a crucial role in preventing us from falling when we lose our balance. However, to recover balance successfully, the central nervous system has to be able to control the stepping or grasping movement to deal with "environmental constraints" (i.e. objects and architectural features that can obstruct stepping or serve as handholds to grasp), and hence must somehow monitor the location of potential constraints as we move about in our daily lives. The need to monitor these environmental features suggests a critical role for visual attention, gaze control, and spatial memory, all of which are known to decline with aging. Although no studies have examined the effects on balance control, it is known that such deficits can impair other motor behaviors such as driving and can be successfully countered using a computer-based "visual training" intervention designed to improve the ability to rapidly extract information from the peripheral visual field (the so-called "Useful Field of View", or UFOV).

The proposed research will use an analogous approach to improve balance control. Specifically, we will test whether: 1) the UFOV® computer-based visual-training program or a commercially available video game leads to improved ability to use peripheral vision to monitor changes in the spatial features of the surrounding environment, and 2) whether such changes in visual processing are associated with improved ability to rapidly reach and grasp a handrail for support, in response to a sudden unpredictable balance perturbation. Older adults with documented deficits in UFOV scores will be randomly assigned to either the visual training (UFOV or video game) or a control group. Each training group will undergo two one-hour sessions per week, for five consecutive weeks. Neither group will be given any information as to which training method is expected to be more beneficial.

Participants in the experimental group will complete either the computerized UFOV® speed-of-processing intervention or the video game training intervention. This UFOV intervention focuses on the ability to quickly identify and locate visual targets presented (for brief time intervals) in the central and peripheral visual fields. The training challenges the participant to identify the target(s) in the briefest display duration possible, within increasingly difficult task conditions. Difficulty of the training task is increased by making it more difficult to identify the central target, decreasing the duration of target presentation time, increasing the number of tasks to complete simultaneously, adding distracters, and increasing the eccentricity (visual angle) of the peripheral targets.

Participants in the video game training group will participate in game play sessions using a cartoon-based action video game with increasing levels of challenge and difficulty.

Participants in the control group will complete timed computerized word puzzles during the training sessions. This cognitive task involves levels of social interaction and computer use similar to the experimental group, but is not expected to yield improvements in ability to rapidly process peripheral visuospatial information.

Balance assessments will be performed immediately before and after completion of the intervention programs. Balance perturbations will be delivered using a large (2x2m) computer-controlled motion platform. Subjects will stand at the center of the platform and a motor-driven moveable handhold system will be mounted to the front wall of the platform. In each trial, the handhold (a 10cm rod) will be controlled to move, intermittently and unpredictably, back and forth along a horizontal axis in the frontal plane, before coming to rest at one of four final locations (corresponding to visual angles of 5, 10, 15, and 20 degrees). The moving platform will deliver a small perturbation a few seconds after the final handhold location is reached. Subjects will be told to grasp the handhold as quickly as possible in response to the platform motion. During each trial, subjects will perform a concurrent visual vigilance task, which requires them to continuously look straight ahead at the center of a computer screen. This task is designed to ensure the subjects rely on peripheral vision to acquire the spatial information needed to direct the hand toward the handhold following the onset of the platform perturbation. The absence of any eye movements toward the grasp location will be confirmed via recordings from a head-mounted eye tracker. A motion-analysis system will be used to determine the speed and accuracy of the grasping reactions.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* Functional mobility (no dependence on mobility aids)
* Impaired visual processing (UFOV divided attention score of 200ms or worse)

Exclusion Criteria:

* Neurological or musculoskeletal disorder
* Cognitive disorder (e.g. dementia)
* Uncorrected visual impairments
* Recurrent dizziness or unsteadiness

Ages: 64 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
ability to use peripheral vision to recover balance by grasping a handhold | within one week of starting and completing the intervention

SECONDARY OUTCOMES:
natural gaze and balance-recovery behavior (in responding to a sudden unpredictable balance perturbation while walking in an unfamiliar environment); clinical balance measures; visual-processing measures | within one week of starting and completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Maki, PhD, PEng, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto; Sandra M McKay, PhD, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Centre for Studies in Aging, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada